CLINICAL TRIAL: NCT00160953
Title: Development of a Prostate Deformation Model to Enable Accurate Registration of Endorectal Coil Magnetic Resonance Images (ERC-MRI) to Reference Treatment Planning CT Images
Brief Title: Endorectal Coil Magnetic Resonance Images (ERC-MRI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Abbott (Industry); Canadian Association of Radiation Oncology (Industry); Uro-Oncologic Radiation Award (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UHN REB 05-0041-C
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Procedure: Endorectal Coil Magnetic Resonance Images

SUMMARY:
When we acquired MR images of the prostate gland using a coil (receiver antenna) inside the rectum, we can see areas with tumour in the prostate gland, and well as details of the anatomy. The coil inside the rectum changes the shape of the prostate gland. In order to use this images to help target radiation therapy to the tumour better, we need to deform the images to the original shape of the prostate gland without the coil. In this study, we will develop a way to deform the images accurately.

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma of the prostate
* patient undergoing dose escalated conformal EBRT
* low or intermediate risk prognostic factors: PSA < or equa to20, gleason score <8, T <T3, N category 0 or X, M category 0 or X
* > or equal to 18 years of age
* ECOG performance status 0 or 1

Exclusion Criteria:

* contraindications to MRI
* bleeding diathesis and anti-coagulative therapy that cannot be temporarily ceased precluding insertion of fiducial markers
* IFB or collagen vascular disease
* previous colorectal surgery
* previous pelvic RT

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The primary aim of this study is to develop a prostate deformation model using the finite element method from anatomic MR images of the prostate gland acquired with and without ERC.

CONTACTS AND LOCATIONS:
Overall Officials: Menard Cynthia, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada